CLINICAL TRIAL: NCT02645981
Title: Efficacy and Safety of Donafenib in Patients With Advanced Hepatocellular Carcinoma: a Controlled,Multicentre,Randomised, Phase 3 Trial
Brief Title: Efficacy and Safety of Donafenib in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZGDH3
Record Dates: First submitted 2015-12-31; First posted 2016-01-05 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-10

CONDITIONS: HCC
Keywords: Donafeinb; Sorafenib; Phase 3; Overall Survival
MeSH Terms: interventions — donafenib; Sorafenib

STUDY DESIGN:
Masking Description: open-label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donafenib (Experimental): Drug:Donafenib; Dose:200mg,bid,po.
  Interventions: Drug: Donafenib
- Sorafenib(Nexavar) (Active Comparator): Drug:Sorafenib; Dose:400mg,bid,po.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Donafenib — Donafenib is an oral multikinase inhibitor with antiproliferative and antiangiogenic effects
  Other Names: CM4307
  Arms: Donafenib
Drug: Sorafenib — Control
  Other Names: Nexavar
  Arms: Sorafenib(Nexavar)

SUMMARY:
Donafenib versus sorafenib for advanced hepatocellular cancer.

DETAILED DESCRIPTION:
This phase 3 study of donafenib, an oral multikinase inhibitor that targets Raf kinase and receptor tyrosine kinases, is to assess efficacy and safety in patients wiht advanced hepatocellular carcinoma (HCC).The study is a randomised,controlled,multicentre study.The controlled drug is sorafenib(Nexavar).The primary endpoint is overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old;
* Patients with measurable, histologically or clinical proven, inoperable HCC;
* Patients wtih measurable lesion and proved by independent radiology committee(IRC);
* Child-Pugh (CP) score of 7 or less；
* Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less;
* Patients had not received prior systemic treatments for HCC;
* Life expectancy at least 3 months;
* Adequate hepatic and renal function;
* Adequate hematologic function (platelet count,≥75×109per liter;hemoglobin ≥9.0g per deciliter;neutrophil≥1.5×109per liter,);
* Prothrombin time international normal.

Exclusion Criteria:

* Patients received operate in 3 months;
* Patients received transcatheter arterial chemoembolization（TACE） in 4 weeks;
* Patients had received systemic therapy;
* Patients had prior treatment with sorafenib;
* Central nervous system(CNS) involvement;
* Severe or mild-degree ascitic fluid;
* Main portal vein tumor thrombus;
* Inferior venae cava tumor thrombus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Actual)
Dates: Start 2016-03; Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  Patient visits are scheduled every 8 weeks to monitor efficacy.

SECONDARY OUTCOMES:
Progress Free Survival | 2 years
  Patient visits are scheduled every 8 weeks to monitor efficacy.Progressive disease is measured from the date of randomization until dead or disease progression according to Response Evaluation Criteria in Solid Tumors(Version 1.1)
Percentage of adverse events | 3 years
  Patient visits are scheduled every 4 weeks to monitor safety and drug accountability. Patients were monitored for adverse events by use of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCICTCAE) version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, MD, Study Chair — The PLA 81 Hospital; Feng Bi, MD, Study Chair — West China Hospital
Locations (2):
- China (2):
  - The PLA 81 Hospital, Nanjing, Jiangsu
  - West China Hospital Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bi F, Qin S, Gu S, Bai Y, Chen Z, Wang Z, Ying J, Lu Y, Meng Z, Pan H, Yang P, Zhang H, Chen X, Xu A, Cui C, Zhu B, Wu J, Xin X, Wang J, Shan J, Chen J, Zheng Z, Xu L, Wen X, You Z, Ren Z, Xu J, Du C, Fan Q, Zhang L, Tao M, Jiang D, Wang S, Chen Y, Sheng J, Zhuang X, Wu J. Analysis of common treatment-related adverse events of donafenib and its correlation with efficacy: exploratory analysis of the ZGDH3 study. Eur J Med Res. 2025 Oct 29;30(1):1040. doi: 10.1186/s40001-025-03297-6. PMID 41163129